CLINICAL TRIAL: NCT07222098
Title: An Open-Label, 2-Period, Crossover Study to Evaluate the Effects of a Single Dose of MK-1084 on the Single-Dose Pharmacokinetics of Rosuvastatin and Metformin in Healthy Participants
Brief Title: A Clinical Study of Calderasib (MK-1084) With Rosuvastatin and Metformin in Healthy People (MK-1084-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1084-016; MK-1084-016 (Other: MSD)
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin + metformin (Experimental): Participants will receive rosuvastatin plus metformin
  Interventions: Drug: Rosuvastatin; Drug: Metformin
- Rosuvastatin + metformin + Calderasib (Experimental): Participants will receive rosuvastatin plus metformin plus calderasib
  Interventions: Drug: Rosuvastatin; Drug: Metformin; Drug: Calderasib

INTERVENTIONS:
Drug: Rosuvastatin — Oral tablet
Drug: Metformin — Oral tablet
Drug: Calderasib — Oral tablet
  Other Names: MK-1084
  Arms: Rosuvastatin + metformin + Calderasib

SUMMARY:
Researchers want to learn about calderasib when given with rosuvastatin and metformin in healthy people. The goal of this study is to compare the amount of rosuvastatin and metformin in a person's body over time when given with and without calderasib

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Has body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has history of cancer (malignancy)
* Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-11-19 (Actual); Primary Completion 2025-12-14 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 120 hours post-dose
  Blood samples will be collected at multiple time points to determine the AUC0-inf of rosuvastatin
Maximum Plasma Concentration (Cmax) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 120 hours post-dose
  Blood samples will be collected at multiple time points to determine the Cmax of rosuvastatin
AUC0-inf of Metformin | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to determine the AUC0-inf of metformin

SECONDARY OUTCOMES:
Area Under the Curve From Time 0 to Last Quantifiable Sample (AUC0-last) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 120 hours post-dose
  Blood samples will be collected at multiple time points to determine the AUC0-last of rosuvastatin
Area Under the Curve From Time 0 to 24 Hours (AUC0-24hrs) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 24 hours post-dose
  Blood samples will be collected at multiple time points to estimate AUC0-24
Time to Maximum Plasma Concentration (Tmax) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 120 hours post-dose
  Blood samples will be collected at multiple time points to estimate Tmax
Day 1: Apparent Terminal Half-life (t1/2) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 120 hours post-dose
  Blood samples will be collected at multiple time points to estimate t1/2
Apparent Clearance (CL/F) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 120 hours post-dose
  Blood samples will be collected at multiple time points to estimate CL/F
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Rosuvastatin | Day 1: Predose and at designated timepoints up to 120 hours post-dose
  Blood samples will be collected at multiple time points to estimate Vz/F
AUC0-last of Metformin | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate AUC0-last
AUC0-24hrs of Metformin | Day 1: Predose and at designated timepoints up to 24 hours post-dose
  Blood samples will be collected at multiple time points to estimate AUC0-24
Cmax of Metformin | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate Cmax
Tmax of Metformin | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate Tmax
t1/2 of Metformin | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate t1/2
CL/F of Metformin | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate CL/F
Vz/F of Metformin | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate Vz/F
AUC0-inf of Calderasib | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate AUC0-inf
AUC0-last of Calderasib | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate AUC0-last
AUC0-24hrs of Calderasib | Day 1: Predose and at designated timepoints up to 24 hours post-dose
  Blood samples will be collected at multiple time points to estimate AUC0-24
Cmax of Calderasib | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate Cmax
Plasma Concentration at 24 Hours (C24) of Calderasib | 24 hours post-dose
  Blood samples will be collected to estimate C24
Tmax of Calderasib | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate Tmax
t1/2 of Calderasib | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate t1/2
CL/F of Calderasib | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate CL/F
Vz/F of Calderasib | Day 1: Predose and at designated timepoints up to 72 hours post-dose
  Blood samples will be collected at multiple time points to estimate Vz/F
Amount of Metformin Excreted Unchanged in Urine (Ae) | Day 1: Predose and at designated timepoints up to 48 hours post-dose
  Urine samples will be collected at multiple time points to estimate Ae
Fraction of Metformin Excreted Unchanged in Urine (Fe) | Day 1: Predose and at designated timepoints up to 48 hours post-dose
  Urine samples will be collected at multiple time points to estimate Fe
Renal Clearance of Metformin (CLr) | Day 1: Predose and at designated timepoints up to 48 hours post-dose
  Urine samples will be collected at multiple time points to estimate CLr
Number of Participants Who Experience an Adverse Avent (AE) | Up to approximately 28 days after first dose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced an AE is reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 14 days after first dose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinued study treatment due to an AE is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/